CLINICAL TRIAL: NCT03241121
Title: Study of Eating Patterns with a Smartphone App and the Metabolic Effects of Time Restricted Feeding (TRF) in the Metabolic Syndrome - an Open-label Randomized Controlled Trial of TRF Vs Regular Dietary Advices
Brief Title: Study of Eating Patterns with a Smartphone App and the Effects of Time Restricted Feeding in the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Tinh-Hai Collet, MD, Principal Investigator, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00487; PZ00P3-167826 (Other Grant/Funding Number: Swiss National Science Foundation); SSED-YI 2017 (Other Grant/Funding Number: Swiss Society of Endocrinology and Diabetes)
Record Dates: First submitted 2017-04-02; First posted 2017-08-07 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-08

CONDITIONS: Eating Behavior; Metabolic Syndrome; Obesity; Dyslipidemias; Glucose Intolerance; Steatosis of Liver
Keywords: Time Restricted Feeding; Eating patterns
MeSH Terms: conditions — Feeding Behavior; Metabolic Syndrome; Obesity; Dyslipidemias; Glucose Intolerance; Fatty Liver; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Study Part 1: Prospective longitudinal observational study. Study Part 2/3: Open-label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Time restricted feeding (Experimental): For those in the intervention phase (Part 2)
  Interventions: Behavioral: Time restricted feeding; Device: Eating patterns
- Regular dietary advices (Active Comparator): For those in the intervention phase (Part 2)
  Interventions: Behavioral: Regular dietary advices; Device: Eating patterns

INTERVENTIONS:
Behavioral: Time restricted feeding — To eat only during a self-selected window of 12 hours, with no advice on nutrition quality, quantity or caloric intake
  Arms: Time restricted feeding
Behavioral: Regular dietary advices — Regular dietary advices by a trained dietitian or research nurse according to current nutrition guidelines
  Arms: Regular dietary advices
Device: Eating patterns — Data collection on eating patterns via the smartphone app

SUMMARY:
SwissChronoFood - Study of eating patterns with a smartphone app and the metabolic effects of time restricted feeding in metabolic syndrome

The purpose of this study is to assess eating patterns among teenagers and adults with a new method, going beyond the pen-and-paper food diaries, and to investigate whether time restricted feeding leads to weight loss, improvement in lipid and glucose metabolism in individuals with components of the metabolic syndrome

DETAILED DESCRIPTION:
The prevalence of the metabolic syndrome (MS) is increasing worldwide, due to the progression of its different components (central obesity, elevated blood pressure, impaired glucose tolerance and dyslipidemia), as well as the often associated liver steatosis. One way to tackle the obesity epidemic is to intervene early at the onset in childhood and teenage years - before cardio-metabolic complications have occurred. However, lifestyle programs targeting this age group had limited success in the current obesogenic environment. In particular, weight loss is a key factor in controlling all MS components, yet it is difficult to maintain over time.

Time restricted feeding (TRF) is an approach that emphasizes energy intake limited to certain windows of time within the 24-hour cycle without restrictions on calories or macronutrients. This has emerged as an appealing approach to reduce body weight while improving lipid profile and glucose metabolism. However, TRF has been mostly studied in animals and long-term prospective data on its efficacy and mechanisms in humans is lacking.

Prior to the intervention, the investigators will assess the eating patterns of participants with an innovative smartphone application ('app') which is less intrusive and more reliable than food diaries/questionnaires to assess eating behavior and patterns.

In this project, the investigators will assess eating patterns among teenagers and adults, and investigate whether a controlled TRF intervention leads to beneficial changes in MS components. Study Part 1 uses an epidemiological approach to establish baseline daily eating behavior, physical activity patterns and sleeping habits over 2 weeks (teenagers) and 4 weeks (adults) using the smartphone app. Those individuals meeting criteria for at least one component of MS and who have eaten for >14 hours per 24-hour cycle will be recruited for Study Part 2. In Part 2, participants will be assigned to TRF or active control groups, and followed in this pragmatic randomized controlled trial for 6 weeks (teenagers) and 6 months (adults) to assess the change in their weight and MS components, as well as liver fat deposits. Study Part 3 will investigate the underlying mechanisms of improved metabolic profile with TRF.

ELIGIBILITY:
Key inclusion criteria for both observation and intervention phases (Part 1+2):

* Age ≥ 12 years
* Body mass index ≥ 20 kg/m2 and stable weight (previous 3 months) in adults; BMI ≥ 25th percentile in teenagers
* Smartphone compatible with the app (iOS or Android systems)

Additional inclusion criteria for the intervention phase (Part 2):

* Any component of the metabolic syndrome following the International Diabetes Federation consensus definition
* Eating duration >14h during the observation phase

Additional inclusion criteria for the mechanistic study (Part 3):

* Age 18-40 years, men and pre-menopausal women
* BMI 30-40 kg/m2
* In the fasting state (at least 8 hours)

Key exclusion criteria for both observation and intervention phases (Part 1+2):

* Pregnant and breastfeeding women, plans for maternity during the study
* Major illness/fever over the previous month, active cancer
* Eating disorder, on a diet / weight management, prior bariatric surgery
* Major mental illness, unable to give informed consent
* Current shift work or travel abroad planned in the next month

Additional exclusion criteria for the intervention phase (Part 2):

* Prior cardiovascular event
* Major liver, gastrointestinal, renal or endocrine disorder, diabetes mellitus with hypoglycemic drug(s)
* Major sleep disorder, centrally acting medication
* Lipid lowering drug, hypoglycemic drug, medication affecting the gut

Additional exclusion criteria for the mechanistic study (Part 3):

* Impaired glucose tolerance (pre-diabetes) or diabetes mellitus
* Positive pregnancy test

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Eating duration | From baseline visit to end of observation phase (Part 1: 4 weeks for adults, 2 weeks for teenagers)
  Duration from the first to last caloric intake over 24-hour cycle, collected via the smartphone app.
  Note: Key inclusion criterion for the intervention phase (Part 2).
Change of metabolic syndrome components | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Number of participants with changes in weight and/or lipid profile and/or glucose metabolism in the intervention phase (Part 2).
  Note: Changes of the different components will be analyzed separately as secondary outcomes.

SECONDARY OUTCOMES:
Adherence to TRF intervention | From randomization visit to close-out visit (Part 2: 6 months for adults, 6 weeks for teenagers)
  After allocation to the TRF arm, assessment of the adherence to the intervention, as measured by eating duration from the first to last caloric intake over 24-hour cycle.
Weight change | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Part of the composite primary outcome in the intervention phase (Part 2)
Change in lipid profile | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Part of the composite primary outcome in the intervention phase (Part 2)
Change in glucose metabolism | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Part of the composite primary outcome in the intervention phase (Part 2)
Change in blood pressure | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Systolic and diastolic blood pressure
Change in hepatic steatosis / fibrosis score | From randomization visit to close-out visit (Part 2: 6 months for adults, 6 weeks for teenagers)
  As measured by the Fibroscan device
Change in number of meals per day | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Temporal analysis of caloric intake events collected by the smartphone app
Change in meal intervals | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Temporal analysis of caloric intake events collected by the smartphone app
Change in fraction of calories consumed after noon | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Estimation of caloric content from food pictures collected by the smartphone app
Change in fraction of calories consumed after 6pm | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Estimation of caloric content from food pictures collected by the smartphone app
Change in eating pattern difference between weekdays and weekends | From baseline visit to close-out visit (Part 1: 4 weeks for adults, 2 weeks for teenagers; followed by Part 2: 6 months for adults, 6 weeks for teenagers)
  Indirect assessment of different lifestyle habits during weekdays and weekends

OTHER OUTCOMES:
Change in fat mass | From randomization visit to close-out visit (Part 3: 6 months, only adults)
  Body composition as measured by dual energy X-ray absorptiometry (DEXA)
Change in fat free mass | From randomization visit to close-out visit (Part 3: 6 months, only adults)
  Body composition as measured by dual energy X-ray absorptiometry (DEXA)
Change in diurnal rhythms of cortisol secretion | From randomization visit to close-out visit (Part 3: 6 months, only adults)
  Repeated measurements of cortisol over a 24-hour cycle
Change in diurnal rhythms of melatonin secretion | From randomization visit to close-out visit (Part 3: 6 months, only adults)
  Repeated measurements of melatonin over a 24-hour cycle
Change in physical activity | From randomization visit to close-out visit (Part 3: 6 months, only adults)
  As measured by actigraphy
Change in sleep/wake cycles | From randomization visit to close-out visit (Part 3: 6 months, only adults)
  As measured by actigraphy
Eating duration - alternative definition of the primary outcome | From baseline visit to end of observation phase (Part 1: 4 weeks for adults, 2 weeks for teenagers)
  Alternative definition of eating duration accounting for 2.5-97.5th percentiles of caloric intake over 24 hours, presumably less sensitive to the occasionally forgotten food picture event

CONTACTS AND LOCATIONS:
Overall Officials: Tinh-Hai Collet, MD, Principal Investigator — University of Lausanne Hospitals
Locations (2):
- Switzerland (2):
  - Inselspital, Klinik für Allgemeine Innere Medizin, Bern, Canton of Bern
  - University Hospital of Lausanne (CHUV), Lausanne

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset of selected variables that underlie results in a publication. Some data may not be amenable to complete anonymization and will not be shared to ensure appropriate confidentiality of participant's data.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Upon appropriate data request by other scientists

REFERENCES:
- [Background] Buso G, Favre L, Vionnet N, Gonzalez-Rodriguez E, Hans D, Puder JJ, Dubath C, Eap CB, Raffoul W, Collet TH, Mazzolai L. Body Composition Assessment by Dual-Energy X-Ray Absorptiometry: A Useful Tool for the Diagnosis of Lipedema. Obes Facts. 2022;15(6):762-773. doi: 10.1159/000527138. Epub 2022 Oct 28. PMID 36310013
- [Background] Phillips NE, Mareschal J, Schwab N, Manoogian ENC, Borloz S, Ostinelli G, Gauthier-Jaques A, Umwali S, Gonzalez Rodriguez E, Aeberli D, Hans D, Panda S, Rodondi N, Naef F, Collet TH. The Effects of Time-Restricted Eating versus Standard Dietary Advice on Weight, Metabolic Health and the Consumption of Processed Food: A Pragmatic Randomised Controlled Trial in Community-Based Adults. Nutrients. 2021 Mar 23;13(3):1042. doi: 10.3390/nu13031042. PMID 33807102
- [Background] Borloz S, Bucher Della Torre S, Collet TH, Jotterand Chaparro C. Consumption of Ultraprocessed Foods in a Sample of Adolescents With Obesity and Its Association With the Food Educational Style of Their Parent: Observational Study. JMIR Pediatr Parent. 2021 Nov 15;4(4):e28608. doi: 10.2196/28608. PMID 34779776
- [Background] Papageorgiou M, Biver E, Mareschal J, Phillips NE, Hemmer A, Biolley E, Schwab N, Manoogian ENC, Gonzalez Rodriguez E, Aeberli D, Hans D, Pot C, Panda S, Rodondi N, Ferrari SL, Collet TH. The effects of time-restricted eating and weight loss on bone metabolism and health: a 6-month randomized controlled trial. Obesity (Silver Spring). 2023 Feb;31 Suppl 1(Suppl 1):85-95. doi: 10.1002/oby.23577. Epub 2022 Oct 14. PMID 36239695